CLINICAL TRIAL: NCT03370120
Title: An Open-Label, Multicenter, Extension Study to Evaluate the Safety and Efficacy of Padsevonil as Adjunctive Treatment of Focal-Onset Seizures in Adult Subjects With Drug-Resistant Epilepsy
Brief Title: Study to Test the Safety and Efficacy of Padsevonil as Adjunctive Treatment of Focal-onset Seizures in Adult Subjects With Drug-resistant Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizure
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0093; 2017-003241-26 (EudraCT Number)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Drug-Resistant Epilepsy; Focal-Onset Seizures
Keywords: Drug-Resistant Epilepsy; Padsevonil
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures | interventions — padsevonil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Padsevonil (Experimental): Padsevonil will be administered in an open-label manner. The individual starting dose of each subject will be the one at the end of the parent study.
  Once subjects enter EP0093 further individual dose adjustments are allowed after 1 week to the extent possible with the combination of tablet strengths available.
  Interventions: Drug: Padsevonil

INTERVENTIONS:
Drug: Padsevonil — * Pharmaceutical Form: film-coated tablet
  * Route of Administration: Oral use

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability of Padsevonil administered at individualized doses as adjunctive treatment for subjects with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult (18 years of age or more )
* Subject with epilepsy who has completed 1 of the previous Padsevonil (PSL) studies which allow access to the present study
* Female subjects of child bearing potential must have a serum negative pregnancy test at the Entry Visit, which is confirmed to be negative by urine testing prior to further dispensing at each study visit thereafter. Subjects will be withdrawn from the study as soon as pregnancy is known. Female subjects will use an efficient form of contraception for the duration of the study and for a period of 3 months after their final dose of PSL.

Exclusion Criteria:

* Subject has any severe medical, neurological, or psychiatric condition, or laboratory value which may have an impact on the safety of the subject
* Subject has active suicidal ideation as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the 'Since Last Visit' version of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Subject has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (>= l.5x ULN total bilirubin if known Gilbert's syndrome) at the Entry Visit
* Subject has a clinically-significant abnormality on electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Subject has an abnormality on echocardiogram at last echocardiogram assessment, or foreseen in parent study as assessed by central reader that is accompanied by clinical symptoms or a Grade 2* (or higher)/moderate severity abnormality, or a history of rheumatic heart disease, or other known valvular abnormalities (*according to the ASE Guidelines, 2017; Zoghbi et al 2017)
* Female subject who plans to be pregnant or is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (156):
- United States (25):
  - Ep0093 839, Chandler, Arizona
  - Ep0093 815, La Jolla, California
  - Ep0093 801, San Francisco, California
  - Ep0093 803, Honolulu, Hawaii
  - Ep0093 638, Fort Wayne, Indiana
  - Ep0093 707, Lexington, Kentucky
  - Ep0093 822, Baltimore, Maryland
  - Ep0093 818, Bethesda, Maryland
  - Ep0093 889, Boston, Massachusetts
  - Ep0093 645, Golden Valley, Minnesota
  - Ep0093 817, Saint Paul, Minnesota
  - Ep0093 806, Hackensack, New Jersey
  - Ep0093 893, Syracuse, New York
  - Ep0093 895, The Bronx, New York
  - Ep0093 890, Chapel Hill, North Carolina
  - Ep0093 884, Charlotte, North Carolina
  - Ep0093 642, Columbia, Ohio
  - Ep0093 802, Philadelphia, Pennsylvania
  - Ep0093 838, Cordova, Tennessee
  - Ep0093 835, Nashville, Tennessee
  - Ep0093 805, Austin, Texas
  - Ep0093 844, Austin, Texas
  - Ep0093 824, Round Rock, Texas
  - Ep0093 870, San Antonio, Texas
  - Ep0093 639, Renton, Washington
- Australia (8):
  - Ep0093 855, Box Hill
  - Ep0093 857, Clayton
  - Ep0093 850, Fitzroy
  - Ep0093 853, Heidelberg
  - Ep0093 859, Herston
  - Ep0093 852, Melbourne
  - Ep0093 856, Randwick
  - Ep0093 854, Westmead
- Belgium (5):
  - Ep0093 102, Bruges
  - Ep0093 101, Brussels
  - Ep0093 105, Ghent
  - Ep0093 100, Leuven
  - Ep0093 107, Ottignies
- Bosnia and Herzegovina (2):
  - Ep0093 075, Sarajevo
  - Ep0093 082, Tuzla
- Bulgaria (7):
  - Ep0093 150, Blagoevgrad
  - Ep0093 151, Pleven
  - Ep0093 153, Pleven
  - Ep0093 156, Pleven
  - Ep0093 152, Sofia
  - Ep0093 154, Sofia
  - Ep0093 155, Sofia
- Canada (3):
  - Ep0093 200, Greenfield Park
  - Ep0093 205, London
  - Ep0093 201, Montreal
- Ep0093 125, Zagreb, Croatia
- Czechia (5):
  - Ep0093 254, Brno
  - Ep0093 255, Ostrava
  - Ep0093 250, Prague
  - Ep0093 251, Prague
  - Ep0093 253, Prague
- Denmark (2):
  - Ep0093 016, Aarhus
  - Ep0093 015, Odense
- Estonia (3):
  - Ep0093 276, Tallinn
  - Ep0093 277, Tallinn
  - Ep0093 275, Tartu
- Ep0093 027, Tampere, Finland
- France (6):
  - Ep0093 307, Clermont-Ferrand
  - Ep0093 309, Dijon
  - Ep0093 300, Lille
  - Ep0093 302, Montpellier
  - Ep0093 303, Rennes
  - Ep0093 301, Strasbourg
- Germany (14):
  - Ep0093 365, Berlin
  - Ep0093 362, Bernau
  - Ep0093 363, Bielefeld
  - Ep0093 358, Bonn
  - Ep0093 350, Frankfurt
  - Ep0093 360, Freiburg im Breisgau
  - Ep0093 368, Jena
  - Ep0093 366, Kehl
  - Ep0093 357, Leipzig
  - Ep0093 353, Marburg
  - Ep0093 354, München
  - Ep0093 351, Münster
  - Ep0093 356, Osnabrück
  - Ep0093 352, Tübingen
- Greece (2):
  - Ep0093 426, Thessaloniki
  - Ep0093 427, Thessaloniki
- Hungary (3):
  - Ep0093 400, Budapest
  - Ep0093 403, Budapest
  - Ep0093 402, Debrecen
- Ep0093 035, Cork, Ireland
- Italy (10):
  - Ep0093 462, Bologna
  - Ep0093 450, Cagliari
  - Ep0093 451, Foggia
  - Ep0093 461, Foggia
  - Ep0093 452, Milan
  - Ep0093 459, Pavia
  - Ep0093 458, Pozzilli
  - Ep0093 455, Roma
  - Ep0093 457, Roma
  - Ep0093 460, Roma
- Japan (14):
  - Ep0093 526, Asahikawa
  - Ep0093 501, Asaka
  - Ep0093 521, Bunkyō City
  - Ep0093 511, Fukuoka
  - Ep0093 504, Hamamatsu
  - Ep0093 505, Hiroshima
  - Ep0093 513, Hōfu
  - Ep0093 507, Itami
  - Ep0093 514, Kyoto
  - Ep0093 512, Nagakute
  - Ep0093 510, Niigata
  - Ep0093 515, Saitama
  - Ep0093 509, Shizuoka
  - Ep0093 529, Yonago
- Lithuania (2):
  - Ep0093 703, Kaunas
  - Ep0093 702, Vilnius
- Mexico (2):
  - Ep0093 553, Culiacán
  - Ep0093 552, México
- Poland (12):
  - Ep0093 601, Gdansk
  - Ep0093 607, Grodzisk Mazowiecki
  - Ep0093 605, Katowice
  - Ep0093 616, Katowice
  - Ep0093 603, Krakow
  - Ep0093 614, Krakow
  - Ep0093 604, Lublin
  - Ep0093 610, Lublin
  - Ep0093 606, Nowa Sól
  - Ep0093 600, Poznan
  - Ep0093 609, Poznan
  - Ep0093 602, Świdnik
- Ep0093 926, Bucharest, Romania
- Ep0093 327, Belgrade, Serbia
- Ep0093 004, Bardejov, Slovakia
- Spain (15):
  - Ep0093 662, Alicante
  - Ep0093 668, Barakaldo
  - Ep0093 651, Barcelona
  - Ep0093 652, Barcelona
  - Ep0093 664, Barcelona
  - Ep0093 666, Córdoba
  - Ep0093 658, L'Hospitalet de Llobregat
  - Ep0093 656, Madrid
  - Ep0093 660, Madrid
  - Ep0093 667, Madrid
  - Ep0093 674, Madrid
  - Ep0093 659, Málaga
  - Ep0093 665, Terrassa
  - Ep0093 657, Valencia
  - Ep0093 653, Valladolid
- Turkey (Türkiye) (5):
  - Ep0093 900, Istanbul
  - Ep0093 901, Istanbul
  - Ep0093 904, Istanbul
  - Ep0093 906, Istanbul
  - Ep0093 909, Istanbul
- United Kingdom (5):
  - Ep0093 752, Birmingham
  - Ep0093 766, Brighton
  - Ep0093 751, Swansea
  - Ep0093 753, Swansea
  - Ep0093 764, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in August 2018 and concluded in December 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set. Participants who had completed a padsevonil (PSL) parent study (EP0091 [NCT03373383] or EP0092 [NCT03739840]) were enrolled in this study.
Groups:
- Padsevonil: Participants received padsevonil tablets at a dose of 100 milligrams/day (mg/day) to 800 mg/day up to approximately 2 years.
Period: Overall Study
Arm/Group | Padsevonil
Started | 406
Completed | 0
Not Completed | 406
Not completed — Adverse event, non-fatal | 24
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 37
Not completed — Per sponsor's instructions | 1
Not completed — Study was terminated by parent company UCB | 2
Not completed — The study was ended by the promoter | 3
Not completed — Discontinuation of drug development | 3
Not completed — End of project | 2
Not completed — Premature study closure | 2
Not completed — Premature program termination | 1
Not completed — Premature study termination | 7
Not completed — Trial terminated by sponsor | 2
Not completed — Trial discontinued by sponsor | 2
Not completed — Study ended | 15
Not completed — Clinical trial has been cancelled | 1
Not completed — End of study per sponsor decision | 2
Not completed — Promoter's decision | 2
Not completed — The trial has been suspended | 3
Not completed — Sponsor stopped PSL development based on data | 3
Not completed — Early termination by order of sponsor | 2
Not completed — Discontinuation of the study | 5
Not completed — End of clinical trial discontinuation | 1
Not completed — Because the clinical trial ended halfway | 4
Not completed — Development discontinued | 5
Not completed — Padsenovil program closed | 3
Not completed — End of project | 2
Not completed — Termination of project | 1
Not completed — The study was interrupted by sponsor | 4
Not completed — The protocol was interrupted by sponsor | 1
Not completed — End of sponsor decision | 1
Not completed — The study was terminated prematurely by study lead | 1
Not completed — Early termination of studies | 5
Not completed — This study is ended early | 1
Not completed — End of padsevonil program | 2
Not completed — Decision of sponsor | 6
Not completed — Asked by the sponsor | 3
Not completed — Sponsor decision to stop the protocol | 1
Not completed — PI decision poor compliance from participant | 1
Not completed — Promoter ended the study | 3
Not completed — Premature study close by sponsor's decision | 4
Not completed — Study terminated by sponsor | 33
Not completed — Sponsor prematurely terminated this study | 2
Not completed — Sponsor decision to terminate study | 63
Not completed — Program closure | 3
Not completed — Study ended prematurely | 1
Not completed — Study stopped by sponsor | 2
Not completed — Program termination | 55
Not completed — Sponsor decision | 62
Not completed — Sponsor study closure | 10

BASELINE CHARACTERISTICS:
Population: The Safety Set (SS) consisted of all enrolled participants who were administered at least 1 dose of PSL, based on the first dose date from the first administration of study medication Case Report form (CRF).
Groups:
- Padsevonil: Participants received PSL tablets at a dose of 100 mg/day to 800 mg/day up to approximately 2 years.
Arm/Group | Padsevonil
Number analyzed (Participants) | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 395
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231
  Male | 175
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaskan native | 5
  Asian | 38
  Black | 6
  Native Hawaiian or other Pacific Islander | 5
  White | 343
  Other/mixed | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Reported by the Participant and/or Caregiver or Observed by the Investigator During the Entire Study
Description: An Adverse Event is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE was defined as any event that was not present prior to the initiation of the first dose of study treatment in this study or any unresolved event already present before initiation of the first dose that worsens in intensity following exposure to the treatment.
Time Frame: From Entry Visit (Week 0) until the Safety Follow-up Visit (up to approximately 2 years)
Population: The Safety Set (SS) consisted of all enrolled participants who were administered at least 1 dose of PSL, based on the first dose date from the first administration of study medication CRF.
Measure: Number; unit: percentage of participants
Groups:
- Padsevonil (SS): Participants received PSL tablets at a dose of 100 mg/day to 800 mg/day up to approximately 2 years. Participants formed the Safety Set (SS).
Arm/Group | Padsevonil (SS)
Number analyzed (Participants) | 406
percentage of participants | 72.2

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal
Description: as for outcome 1
Time Frame: From Entry Visit (Week 0) until the Safety Follow-up Visit (up to approximately 2 years)
Population: The SS consisted of all enrolled participants who were administered at least 1 dose of PSL, based on the first dose date from the first administration of study medication CRF.
Measure: Number; unit: percentage of participants
Groups:
- Padsevonil (SS): Participants received PSL tablets at a dose of 100 mg/day to 800 mg/day up to approximately 2 years. Participants formed the SS.
Arm/Group | Padsevonil (SS)
Number analyzed (Participants) | 406
percentage of participants | 5.2

3. Primary Outcome: Change From Baseline (From the Respective Parent Study [EP0091 or EP0092]) in Observable Focal-onset Seizure Frequency Over the Evaluation Period
Description: Seizure frequency refers to 28-day adjusted frequency. Observable focal-onset seizures refer to Type IAl, IB, and IC (according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures, 1981). Focal-onset seizures include all Type I seizures.
Time Frame: From Baseline in respective parent study over the Evaluation Period (up to approximately 2 years) in this study
Population: Full Analysis Set (FAS) consisted of all enrolled participants who were administered at least 1 dose of PSL or a partial dose of PSL and completed at least 1 seizure diary during the Evaluation Period.
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Groups:
- Padsevonil (FAS): Participants received PSL tablets at a dose of 100 mg/day to 800 mg/day up to approximately 2 years. Participants formed the FAS.
Arm/Group | Padsevonil (FAS)
Number analyzed (Participants) | 406
seizures per 28 days | -7.73 (27.52)

ADVERSE EVENTS:
Time Frame: From Entry Visit (Week 0) until the Safety Follow-up Visit (up to approximately 2 years)
Description: A TEAE was defined as any event that was not present prior to the initiation of the first dose of study treatment in this study or any unresolved event already present before initiation of the first dose that worsens in intensity following exposure to the treatment.
Arm/Group | Padsevonil (SS)
All-Cause Mortality (participants affected / at risk) | 0/406
Serious Adverse Events (participants affected / at risk) | 48/406
Other Adverse Events (participants affected / at risk) | 184/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Padsevonil (SS) (N=406)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Mycoplasma test positive (Investigations) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 7 (8)
Focal dyscognitive seizures (Nervous system disorders) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 5 (8)
Migraine (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 2 (3)
Postictal state (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
Seizure cluster (Nervous system disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 5 (5)
Syncope (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Vagal nerve stimulator implantation (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Padsevonil (SS) (N=406)
Somnolence (Nervous system disorders) | 66 (76)
Headache (Nervous system disorders) | 59 (138)
Dizziness (Nervous system disorders) | 43 (63)
Memory impairment (Nervous system disorders) | 21 (38)
Fatigue (General disorders) | 47 (56)
Nasopharyngitis (Infections and infestations) | 29 (42)
Insomnia (Psychiatric disorders) | 23 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03370120/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03370120/SAP_001.pdf